CLINICAL TRIAL: NCT02881567
Title: A Phase 3b, 12-month, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of BIIB019, Daclizumab, in Subjects With Relapsing-Remitting Multiple Sclerosis (RRMS) Switching From Natalizumab (SUSTAIN)
Brief Title: Efficacy and Safety of Daclizumab in Participants With RRMS Switching From Natalizumab
Acronym: SUSTAIN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated in line with Biogen decision to withdraw Zinbryta from the market and not to pursue further studies of daclizumab in MS.
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205MS305; 2016-002820-10 (EudraCT Number)
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Relapsing-Remitting Multiple Sclerosis (RRMS)
Keywords: Multiple Sclerosis; Daclizumab; Tysabri-Switch
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daclizumab (Experimental)
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Daclizumab — High yield formulation
  Other Names: BIIB019; Zinbryta

SUMMARY:
The primary objective of the study is to evaluate the effects of treatment with daclizumab on the proportion of participants relapse-free at 6 months in Relapsing-Remitting Multiple Sclerosis (RRMS) participants, who switched from treatment with natalizumab to daclizumab due to safety concerns. The secondary objectives of this study in this study population are to evaluate the effects of daclizumab on the following: 1) Multiple Sclerosis (MS) relapse activity including the annualized relapse rate (ARR) and the proportion of participants experiencing relapses requiring hospitalization and/or steroid treatment; 2) MS-related outcomes measured using magnetic resonance imaging (MRI); 3) Safety and tolerability in participants previously treated with natalizumab.

ELIGIBILITY:
Key Inclusion Criteria

* Must have documented diagnosis of RRMS (McDonald 2010 Criteria) at screening [Polman 2011].
* Must have been treated with natalizumab for at least the 12 months prior to screening and have not missed 2 or more consecutive scheduled doses.
* Must be naïve to daclizumab and other forms of daclizumab such as Zenapax® prior to enrollment.
* Must have a confirmed Expanded Disability Status Scale (EDSS) score of 0 to 5.5, inclusive, at screening.
* Female participants of childbearing potential must practice effective contraception from Day -1 and be willing and able to continue contraception for duration of the study.

Key Exclusion Criteria

* Current participation in another investigational study.
* Diagnosis of primary progressive, secondary progressive, or progressive relapsing MS (as defined by Lublin and Reingold) [Lublin 2014].
* Females breastfeeding, pregnant, or planning to become pregnant; or women who have a positive pregnancy test result during screening.
* History of drug or alcohol abuse (as defined by the Investigator) within 1 year prior to screening.
* History of severe hypersensitivity (e.g., anaphylaxis or anaphylactoid reactions) to the active ingredient or any of the excipients.
* History of severe opportunistic infections (including progressive multifocal leukoencephalopathy (PML)) or any clinically significant, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (other than MS), dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
* Discontinued natalizumab due to suspicion of PML.
* Known active malignancies (participants with cutaneous basal cell carcinoma that has been completely excised prior to study entry remain eligible).
* The participant is using another MS therapy concomitantly.
* Known history of human immunodeficiency virus (HIV).
* Positive test result for Hepatitis C virus (test for hepatitis C virus antibody [HCV Ab]) or hepatitis B virus (test for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb]).
* The participant has been treated with immunosuppressive or immunomodulating treatments including mitoxantrone, azathioprine, methotrexate, cyclophosphamide, or mycophenolate mofetil.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- United States (3):
  - Research Site, Tampa, Florida
  - Research Site, Des Moines, Iowa
  - Research Site, Milwaukee, Wisconsin
- Research Site, Edmonton, Alberta, Canada
- Germany (4):
  - Research Site, Munich, Bavaria
  - Research Site, Potsdam, Brandenburg
  - Research Site, Dresden, Saxony
  - Research Site, Hamburg
- Italy (2):
  - Research Site, Pozzilli, Isernia
  - Research Site, Napoli
- Research Site, Guaynabo, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled in the study at 11 investigative sites in Canada, Germany, Italy, and the United States from 05 April 2017 to 12 September 2018.
Pre-assignment Details: Participants who discontinued treatment with natalizumab due to safety concerns were enrolled to receive daclizumab 150 milligrams (mg) per 1.0 milliliter (mL).
Groups:
- Daclizumab: Participants previously treated with natalizumab for at least 12 months and who discontinued treatment, received daclizumab 150 mg per 1.0 mL administered subcutaneously once a month for up to 11 months.
Period: Overall Study
Arm/Group | Daclizumab
Started | 41
Completed | 23
Not Completed | 18
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3
Not completed — Consent withdrawn | 1
Not completed — Investigator decision | 1
Not completed — Study terminated by sponsor | 9
Not completed — Reason not Specified | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants enrolled in the study.
Arm/Group | Daclizumab
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9
  Black or African American | 4
  Not Reported Due to Confidentiality Regulation | 27
  Other (Aboriginal) | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Relapse-free at Month 6
Description: Relapses were defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Examining Neurologist. The Kaplan-Meier estimate of the percentage of participants relapse-free at Month 6 is reported.
Time Frame: Month 6
Population: FAS included all participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Daclizumab
Number analyzed (Participants) | 41
percentage of participants | 66.615

2. Secondary Outcome: Percentage of Participants Relapse-free at Month 12
Description: Relapses were defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Examining Neurologist.
Time Frame: Month 12
Population: The study was terminated. No participants reached the 12-month time point.
Arm/Group | Daclizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Experiencing Relapse Requiring Hospitalization and/or Steroid Treatment at Month 12
Description: as for outcome 2
Time Frame: Month 12
Population: The study was terminated. No participants reached the 12-month time point.
Arm/Group | Daclizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Annualized Relapse Rate (ARR) at Month 12
Description: Relapses were defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Examining Neurologist. The ARR was calculated by tabulating the total number of relapses experienced in the group divided by the number of days up to the end of Month 12, and the ratio then multiplied by 365.
Time Frame: Month 12
Population: The study was terminated. No participants reached the 12-month time point.
Arm/Group | Daclizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With New Gadolinium-Enhanced (Gd+) and T1 Hypointense Lesions at Months 6 and 12
Description: New Gadolinium-Enhanced (Gd+) and T1 Hypointense Lesions were assessed using magnetic resonance imaging (MRI).
Time Frame: Months 6 and 12
Population: FAS included all participants enrolled in the study. Number Analyzed is the number of participants with available assessment. No data was collected for T1 Hypointense Lesions at Month 6. No participants reached the 12-month time point since the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Daclizumab
Number analyzed (Participants) | 41
Participants
  Month 6, Gd+ Lesions: number analyzed (Participants) | 11
  Month 6, Gd+ Lesions | 3
  Month 6, T1 Hypointense Lesions: number analyzed (Participants) | 0
  Month 12, Gd+ Lesions: number analyzed (Participants) | 0
  Month 12, T1 Hypointense Lesions: number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With New and Newly Enlarged T2 Hypointense Lesions at Months 6 and 12
Description: New and newly enlarged T2 Hypointense Lesions were measured by MRI.
Time Frame: Months 6 and 12
Population: FAS included all participants enrolled in the study. Number Analyzed is the number of participants with available assessment. No participants reached the 12-month time point since the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Daclizumab
Number analyzed (Participants) | 41
Participants
  Month 6: number analyzed (Participants) | 11
  Month 6 | 3
  Month 12: number analyzed (Participants) | 0

7. Secondary Outcome: Permanent Discontinuation Rate of Daclizumab at Month 12
Description: Permanent Discontinuation Rate was calculated as the ratio of number of participants who had permanently discontinued daclizumab prior to Month 12 over the total number of participants who received at least 1 dose of daclizumab in the study.
Time Frame: Month 12
Population: The study was terminated. No participants reached the 12-month time point.
Arm/Group | Daclizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death or in the view of the Investigator, places the participant at immediate risk of death or requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability or results in a birth defect.
Time Frame: First dose of study drug to within 30 days of last dose (up to 11 months)
Population: Safety Population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Daclizumab
Number analyzed (Participants) | 41
Participants
  Participants with AEs | 27
  Participants with SAEs | 9

9. Secondary Outcome: Number of Participants With Clinically Relevant Shifts in Laboratory Assessments
Description: Clinical Laboratory assessments were tests of Chemistry and Hematology. The investigator determined if any of the laboratory results were clinically relevant shifts from Baseline.
Time Frame: First dose of study drug to within 30 days of last dose (up to 11 months)
Population: Safety Population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Daclizumab
Number analyzed (Participants) | 41
Participants | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 30 days of last dose (up to 11 months)
Arm/Group | Daclizumab
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 9/41
Other Adverse Events (participants affected / at risk) | 23/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclizumab (N=41)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Encephalitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 2
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclizumab (N=41)
Lymphadenopathy (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Injection site pain (General disorders) | 7
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 4
Migraine (Nervous system disorders) | 3
Multiple sclerosis relapse (Nervous system disorders) | 7
Depression (Psychiatric disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02881567/SAP_000.pdf
  • Study Protocol (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT02881567/Prot_001.pdf